CLINICAL TRIAL: NCT02626130
Title: A Pilot Study of Tremelimumab With or Without Tissue Cryoablation in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Tremelimumab With or Without Cryoablation in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0539; NCI-2016-00008 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0539 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-12-04; First posted 2015-12-10 (Estimated); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Clear Cell Renal Cell Carcinoma; Metastatic Renal Cell Cancer; Stage IV Renal Cell Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Cryosurgery; tremelimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (tremelimumab) (Experimental): Patients receive tremelimumab IV over 60 minutes at weeks 1 and 5. Within 4-6 weeks later, patients undergo surgery or biopsy. After surgery or biopsy, patients receive tremelimumab IV Q4W for 3 doses, and then every Q12W in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery; Biological: Tremelimumab
- Arm B (tremelimumab and cryoablation) (Experimental): Patients undergo cryoablation and receive tremelimumab IV over 60 minutes at weeks 1 (2-6 days after cryoablation) and 5. Within 4-6 weeks later, patients undergo surgery or biopsy. After surgery or biopsy, patients receive tremelimumab IV Q34W for 3 doses, and then Q12W in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Cryosurgery; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery; Biological: Tremelimumab

INTERVENTIONS:
Procedure: Cryosurgery — Undergo cryoablation
  Other Names: cryoablation; cryosurgical ablation
  Arms: Arm B (tremelimumab and cryoablation)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Ticilimumab

SUMMARY:
This randomized pilot clinical trial studies the side effects of tremelimumab with or without tissue cryoablation in treating patients with kidney cancer that has spread to other places in the body. Tremelimumab binds to a protein called cytotoxic T-lymphocyte-associated protein 4 (CTLA-4), which is found on the surface of T cells (a type of white blood cell). Tremelimumab may block CTLA-4 and help the immune system kill cancer cells. Cryoablation is a procedure that uses a hollow, thin tube called a cryoprobe to freeze and destroy cancer tissue. It is not yet known whether tremelimumab with or without cryoablation is effective in treating patients with kidney cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate safety of tremelimumab alone and in combination with cryoablation in patients with metastatic renal cell carcinoma (RCC).

SECONDARY OBJECTIVES:

I. To explore the longitudinal values for immunological variables (including cluster of differentiation [CD]4+ ICOS+ T cells; effector to regulatory T cell ratio; absolute lymphocyte count) following treatment with tremelimumab in patients with metastatic RCC, and evaluate difference between combination cryoablation and tremelimumab in comparison to tremelimumab alone.

II. To determine the objective response rate and progression-free survival of patients treated with tremelimumab with or without cryoablation.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive tremelimumab intravenously (IV) over 60 minutes at weeks 1 and 5. Within 4-6 weeks later, patients undergo surgery or biopsy. After surgery or biopsy, patients receive tremelimumab IV every 4 weeks (Q4W) for 3 doses, and then every 12 weeks (Q12W) in the absence of disease progression or unacceptable toxicity.

ARM B: Patients undergo cryoablation and receive tremelimumab IV over 60 minutes at weeks 1 (2-6 days after cryoablation) and 5. Within 4-6 weeks later, patients undergo surgery or biopsy. After surgery or biopsy, patients receive tremelimumab IV Q4W for 3 doses, and then Q12W in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30, 60, and 90 days, and then every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic renal cell carcinoma (clear cell or non clear cell)

  * One metastatic site amenable to cryoablation
  * Patients with a single metastatic site may be enrolled if that site is amenable to ablation; however these patients will not be counted in secondary measures of response unless there is new disease detected during follow up
  * Eligible for cytoreductive nephrectomy, metastasectomy, or repeated biopsy; biopsy site cannot be lung, mediastinal lymph node, or bone (unless soft tissue component)
* Patients with any number of prior therapies with anti-angiogenic agents or immunotherapy with the exception of any previous anti-CTLA-4 directed agents are allowed; a 2 week washout period is required for all agents, except for bevacizumab where a 4 week washout is required
* Performance status with Eastern Cooperative Oncology Group (ECOG) score =< 2; patients with performance status of 3 may be considered as long as the decline has been of short duration (< 1 month), and is due to their malignancy and not a comorbid condition (example: pain limiting activity)
* Patient's with an International Metastatic Renal Cell Carcinoma Database Consortium (IMDC or Heng) score of 3 or less will be included; score greater than 4 will be excluded; 1 point each: requirement of systemic treatment for metastatic disease less than 1 year of original diagnosis of renal cell carcinoma, a serum calcium greater than 10, anemia, neutrophilia, thrombocytosis, ECOG performance status >= 2
* No history of autoimmune disorders
* White blood cell (WBC) >= 2000/uL
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets >= 75 x 10^3/uL
* Hemoglobin >= 9 g/dL
* Creatinine =< 3 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT) =< 3.0 x ULN for patients without liver metastases; for patients with liver metastasis ALT =< 5 x ULN is allowed
* Bilirubin =< 1.5 x ULN (except for patients with Gilbert's syndrome, who must have a total bilirubin =< 3 mg/dL)
* Ability to understand and willingness to sign a written informed consent document
* Females of childbearing potential who are sexually active with a non-sterilized male partner and non-sterilized males must use a highly effective method of contraception for 28 days prior to the first dose of investigational product, and must agree to continue using such precautions for 180 days after the final dose of investigational product; cessation of contraception after this point should be discussed with a responsible physician; periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception; they must also refrain from egg cell donation for 180 days after the final dose of investigational product; females of childbearing potential are defined as those who are not surgically sterile (ie, bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause); a highly effective method of contraception is defined as one that results in a low failure rate (ie, less than 1% per year) when used consistently and correctly; the acceptable methods of contraception are: barrier method (e.g. male condom with spermicide, copper T intrauterine device, or levonorgestrel-releasing intrauterine system - Mirena) or hormonal methods (e.g. implants, hormone shot or injection, combined pill, minipill, or patch)

Exclusion Criteria:

* Unresolved toxicities from prior anticancer therapy, defined as having not resolved to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03 grade 0 or 1 with the exception of alopecia and laboratory values listed per the inclusion criteria
* Known or suspected autoimmune disease; patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus or autoimmune vasculitis [e.g., Wegener's granulomatosis] are excluded from this study; patients with a history of Hashimoto's thyroiditis only requiring hormone replacement, type I diabetes, or psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are allowed to participate
* Any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first dose of study drug; inhaled steroids and adrenal replacement steroids doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
* Autoimmune disease: patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus or autoimmune vasculitis (e.g., Wegener's granulomatosis) are excluded from this study
* Any underlying medical or psychiatric condition, which in the opinion of the investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events (AEs), such as a condition associated with frequent diarrhea
* Patients with untreated brain metastases
* Major surgery within 4 weeks of enrollment
* History of other malignancies, other than non-melanoma skin cancer, Ta or T1 (low grade) bladder carcinomas, or other low grade cancer of very low clinical impact, unless in complete remission and off therapy for that disease for at least 2 years
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, history of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Untreated symptomatic spinal cord compressions
* Any non-oncology live or attenuated vaccine therapy used for prevention of infectious diseases within 30 days prior to the first dose of tremelimumab; if patients is enrolled, patient should not receive live vaccine during the study and 180 days after the last dose of tremelimumab
* Concomitant therapy with any of the following: interleukin 2 (IL-2), interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids (used in the management of cancer or non-cancer-related illnesses)
* Previous participation in tremelimumab or ipilimumab clinical trial or prior treatment with a CD137 agonist or CTLA-4 inhibitor or agonist
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control from screening to 90 days after the last dose of tremelimumab monotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Up to 2 weeks
  Safety will be recorded through the incidence of adverse events, serious adverse events and specific laboratory abnormalities (worst grade) in each treatment arm. Descriptive statistical analyses will be performed to summarize the incidence of adverse events.
Incidence of extreme toxicities as graded by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 | Up to 2 weeks
  Extreme toxicities will be defined as any grade 3 or higher adverse event that is possibly, probably, or definitely related to therapy that occurs within the first two cycles of therapy with the following exceptions: any grade 3 or higher adverse event that is potentially treatable with steroids will only count as an extreme toxicity if it does not improve to grade 1 or better within 2 weeks of steroid therapy, grade 3 or 4 amylase or lipase abnormalities that are not associated with symptoms or clinical manifestations of pancreatitis, or grade 3 or 4 drug related endocrinopathies which within two weeks of presentation are adequately controlled with only physiologic hormone replacement therapy.

SECONDARY OUTCOMES:
Response rate | Up to 5 years
  Descriptive statistical analyses will be performed to summarize the response rate including summary tables, scatter-plots, box-plots, proportions, 95% credible intervals, median, means, and standard deviations.
Changes in indication markers | Up to 5 years
  Differences of indication markers between arms will be compared using a t-test with transformations of non-normal data, as needed. A mixed model accounting for patient effects will be used to analyze the longitudinal data on immunological values over time.
Progression free survival | Up to 5 years
  Descriptive statistical analyses will be performed.
Longitudinal data on immunological values over time | Up to 13 weeks
  A mixed model accounting for patient effects will be used to analyze the longitudinal data on immunological values over time.

CONTACTS AND LOCATIONS:
Overall Officials: Padmanee Sharma, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Campbell MT, Matin SF, Tam AL, Sheth RA, Ahrar K, Tidwell RS, Rao P, Karam JA, Wood CG, Tannir NM, Jonasch E, Gao J, Zurita AJ, Shah AY, Jindal S, Duan F, Basu S, Chen H, Espejo AB, Allison JP, Yadav SS, Sharma P. Pilot study of Tremelimumab with and without cryoablation in patients with metastatic renal cell carcinoma. Nat Commun. 2021 Nov 4;12(1):6375. doi: 10.1038/s41467-021-26415-4. PMID 34737281
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org